CLINICAL TRIAL: NCT00586157
Title: Efficacy and Safety/Tolerability of Methylphenidate Transdermal System (MTS) for Before-School Dysfunction in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Study of Medication Patch to Treat Children Ages 6-12 With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy Wilens, MD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-P-001633
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; Daytrana; MTS Patch; Methylphenidate Transdermal System
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate Transdermal System (MTS) (Active Comparator)
  Interventions: Drug: Methylphenidate Transdermal System
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — Medication skin patch titrated to 20mg (at 10 mg and 20 mg doses)
  Other Names: Daytrana
  Arms: Methylphenidate Transdermal System (MTS)
Drug: Placebo — Placebo skin patch titrated to 20mg (at 10 mg and 20 mg doses)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effectiveness of a medication skin patch called Methylphenidate Transdermal System (MTS). We will compare the MTS medicated patch to a placebo patch. We want to find out how well it treats ADHD during the early morning hours before a child leaves for school or summertime routines.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 6 to 12 years of age.
* Diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), by DSM-IV, as manifested in clinical evaluation and confirmed by structured interview.
* Participation in structured morning routine (e.g. school, camp, or other organized activities).

Exclusion Criteria:

* Mental retardation (IQ <75).
* Subjects with a medical condition, or treatment that will either jeopardize subject safety or affect the scientific merit of the study.
* Subjects with moderate to severe dermatological atopy.
* Subjects with known structural cardiac abnormalities.
* Organic brain disorders.
* Seizure Disorder.
* Subjects with Tourette's syndrome, or a history of psychosis or bipolar disorder.
* Subjects with current comorbid psychopathology that in the investigator's opinion will warrant immediate treatment or will interfere with the safe execution of the protocol (i.e. Anxiety or Major Depressive Disorder rated as moderate on CGI).
* Subjects with a history of intolerable adverse effects or non-response to methylphenidate.
* Pregnant or nursing females.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilens, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Faraone SV, Hammerness PG, Wilens TE. Reliability and Validity of the Before-School Functioning Scale in Children With ADHD. J Atten Disord. 2018 Sep;22(11):1040-1048. doi: 10.1177/1087054714564623. Epub 2015 Jan 9. PMID 25575616
- [Derived] Wilens TE, Hammerness P, Martelon M, Brodziak K, Utzinger L, Wong P. A controlled trial of the methylphenidate transdermal system on before-school functioning in children with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2010 May;71(5):548-56. doi: 10.4088/JCP.09m05779pur. PMID 20492851

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 subjects signed consent, and 6 discontinued/withdrew consent prior to completing one week of treatment. The remaining 30 subjects were included in data analyses and thus reported.
Groups:
- MTS Then Placebo: MTS in first intervention then Placebo in second intervention
- Placebo Then MTS: Placebo in first intervention then MTS in second intervention
Period: First Intervention
Arm/Group | MTS Then Placebo | Placebo Then MTS
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Worsening behavior | 1 | 0
Period: Second Intervention
Arm/Group | MTS Then Placebo | Placebo Then MTS
Started | 14 | 15
Completed | 12 | 14
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Worsening behavior | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.17 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Attention Deficit Hyperactivity Disorder Rating Scale [Mean (Standard Deviation); unit: Units on a scale] — Units on a scale range from 0-3 on a scale of severity, with 0 being the least severe item score and 3 being the most severe. The possible range of scores for the scale is 0 (least severe) to 54 (most severe).
  Units on a scale | 37.80 (9.08)
Attention Deficit Hyperactivity Disorder Rating Scale - AM [Mean (Standard Deviation); unit: Units on a scale] — Units on a scale range from 0-3 on a scale of severity, with 0 being the least severe item score and 3 being the most severe. The possible range of scores for the scale is 0 (least severe) to 54 (most severe).
  This measure looked at the morning only.
  Units on a scale | 30.83 (11.53)
Before-School Functioning Questionnaire [Mean (Standard Deviation); unit: Units on a Scale] — The questionnaire includes two a sections, a clinician rated 20-item scale and a 14-item self-report section completed collaboratively by child and parent/guardian.
  Units on the clinician rated scale range from 0-3 on a scale of severity, with 0 being the least severe item score and 3 being the most severe. Units on the self-report section ranged from 0-2 on a scale of severity, with 0 being the least severe item score and 2 being the most severe. The possible range of scores for the questionnaire is 88
  Units on a Scale | 40.50 (11.64)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Defined as Change From Baseline on the Investigator Rated DSM-IV Based ADHD Rating Scale, Over the Course of the Day.
Description: Units on a scale range from 0-3 on a scale of severity, with 0 being the least severe item score and 3 being the most severe. The possible range of scores for the scale is 0 (least severe) to 54 (most severe).
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MTS (Drug A) | Placebo
Number analyzed (Participants) | 30 | 29
Units on a scale | 14.76 (14.48) | 28.33 (15.75)
Statistical Analysis 1: Comparison: MTS (Drug A) vs Placebo; Test type: Superiority or Other; p < .001, Z-test

2. Secondary Outcome: Efficacy Defined as Change From Baseline on Investigator and Parental/Self-report Based Rating Scales and Questionnaires
Description: The questionnaire includes two a sections, a clinician rated 20-item scale and a 14-item self-report section completed collaboratively by child and parent/guardian.
  Units on the clinician rated scale range from 0-3 on a scale of severity, with 0 being the least severe item score and 3 being the most severe. Units on the self-report section ranged from 0-2 on a scale of severity, with 0 being the least severe item score and 2 being the most severe. The possible range of scores for the questionnaire is 88
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MTS (Drug A) | Placebo
Number analyzed (Participants) | 30 | 29
Units on a scale | 12.76 (16.65) | 31.37 (17.79)
Statistical Analysis 1: Comparison: MTS (Drug A) vs Placebo; Test type: Superiority or Other; p = .001, Z-test

3. Primary Outcome: Efficacy Defined as Change From Baseline on the Investigator Rated DSM-IV Based ADHD Rating Scale, During the AM.
Description: as for outcome 1
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MTS (Drug A) | Placebo
Number analyzed (Participants) | 30 | 29
Units on a scale | 10.03 (13.18) | 23.22 (14.91)
Statistical Analysis 1: Comparison: MTS (Drug A) vs Placebo; Test type: Superiority or Other; p = .003, Z-test

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | MTS (Drug A) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 26/30 | 7/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTS (Drug A) (N=30) | Placebo (N=29)
Loss of Appetite (General disorders) | 13 | 0
Other (General disorders) | 10 | 3 — MTS (feeling sad, shaky, dizzy; increase in tics/tremors; increase in energy; itchy eyes infected molluscum); PTS (feeling week, shaky, sad; upper respiratory infection)
Gastro-Intestinal (Gastrointestinal disorders) | 9 | 0
Insomnia (General disorders) | 8 | 0
Headaches (General disorders) | 5 | 1
Irritability (General disorders) | 5 | 1
Pruritis at site (Skin and subcutaneous tissue disorders) | 4 | 0
Rhinitis (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No